CLINICAL TRIAL: NCT06103734
Title: AN INTERVENTIONAL EFFICACY AND SAFETY, PHASE 3, DOUBLE-BLIND, 3-ARM, STUDY TO INVESTIGATE PAIN RESPONSE WITH INTRANASAL ZAVEGEPANT COMPARED WITH PLACEBO IN THE ACUTE TREATMENT OF MULTIPLE MIGRAINE ATTACKS IN ADULT PARTICIPANTS
Brief Title: A Study to Learn About Zavegepant as a Treatment for Multiple Migraine Attacks in Adult Participants
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Strategic decision to cancel the study based on adjusted clinical development plan.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: C5301007; 2023-505209-17-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2023-10-06; First posted 2023-10-27 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Migraine
Keywords: CGRP antagonist; zavegepant; intranasal spray
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Intervention Model Description: Randomized by Interactive Web Response System in a 2:1:1 ratio of zavegepant:placebo:placebo stratified by 1)triptan resistant/refractory yes/no 2)stable migraine prophylactic medication yes/no
Who Masked: Participant, Care Provider, Investigator
Masking Description: This is a double-blind study where neither the investigator nor participant will know which arm the participant is assigned (active/placebo).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (3):
- Zavegepant 10 mg (Active Comparator): This is the active arm where the participant will receive 4 doses of the zavegepant 10mg intranasal
  Interventions: Combination Product: Zavegepant 10 mg
- Placebo - Control 1 (Placebo Comparator): This is one of the two placebo arms where the participant will receive 3 doses of placebo and 1 dose of zavegepant 10mg intranasal. Participant will not know which dose will be zavegepant.
  Interventions: Combination Product: Placebo - Control 1
- Placebo - Control 2 (Placebo Comparator): This is one of the two placebo arms where the participant will receive 3 doses of placebo and 1 dose of zavegepant 10mg intranasal. Participant will not know which dose will be zavegepant.
  Interventions: Combination Product: Placebo - Control 2

INTERVENTIONS:
Combination Product: Zavegepant 10 mg — 4 doses of zavegpant 10 mg intranasal spray device
  Arms: Zavegepant 10 mg
Combination Product: Placebo - Control 1 — 3 doses of placebo intranasal spray device and 1 dose of zavegepant 10 mg intranasal spray device
  Arms: Placebo - Control 1
Combination Product: Placebo - Control 2 — 3 doses of placebo intranasal spray device and 1 dose of zavegepant 10 mg intranasal spray device
  Arms: Placebo - Control 2

SUMMARY:
The purpose of this study to show that zavegepant 10 milligrams given through the nose provides:

* freedom from pain, 2 hours after taking the medicine for the first migraine attack.
* consistent freedom from pain, 2 hours after taking the medicine across 4 separate migraine attacks.

This study is seeking participants who:

* are 18 years of age or older.
* have migraine attacks present for at least 1 year with age onset before 50 years old.
* have migraine attacks, on average, lasting about 4 to 72 hours if not treated.
* have 3 to 8 attacks per month but less than15 headache days per month.

If the participant is fit to take part in the study, the participant will receive either the study medicine zavegepant or placebo. A placebo looks like zavegepant but does not contain active ingredients. The study medicine will be given using nasal spray device containing a single amount of zavegepant or matching placebo.

The participants will be instructed to take the study medicine at home if participants have a migraine headache which reaches moderate or severe pain intensity. The participants are expected to treat up to 4 migraines of moderate to severe intensity.

After taking the study medicine, the participant is not allowed to take any other medications for at least 2 hours after taking the study medicine or placebo. Participant can take other medicines after the 2 hours if the migraine is still present. The participant is expected to record on a paper log all medications taken throughout the study.

The study duration is around 26 weeks. This includes a 28-day screening window, up to 20 weeks of treatment period, and a follow up visit at about 4 weeks after taking the study medicine the last time.

The participant is expected to come into the study center up to 4 times. There will be up to 3 telephone contacts including one after taking the study medicine the first time or Month 1 whichever comes first, at Month 3 if the participant is still in the study, and a safety follow-up.

During the study, the participant is expected to complete two sets of questions in an app on a smartphone. This step is done before and after taking the study medicine. The participants must rate:

* Pain
* Pain symptoms
* How the participants are feeling
* General well-being

ELIGIBILITY:
Inclusion Criteria:

1. Participants aged 18 years or older.
2. Participants with minimum 1 year history of migraine with age onset before 50 years of age.

Exclusion Criteria:

1. History of retinal migraine, basilar migraine or hemiplegic migraine.
2. History or current evidence of uncontrolled, unstable or recently diagnosed cardiovascular or cardiometabolic disease.
3. Major depressive disorder or anxiety disorder.
4. Acute or chronic pain syndromes.
5. Conditions that may affect the administration or absorption of the nasal product.
6. History of alcohol abuse and/or illicit drug.
7. Other social, medical, or psychiatric condition that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.
8. Current use of any prohibited concomitant medication(s) or participants unwilling/unable to use a permitted concomitant medication(s)
9. History of use of ergotamine medications or triptans on greater than/equal to 10 days per month on a regular basis for greater than/equal to 3 months. Or history of non-narcotic analgesic intake on greater than/equal to 15 days per month for greater than/equal to 3 months for other pain indications.
10. Participation in clinical trial with non-biological investigational agents or interventional treatments (last study visit occurring) within the 30 days prior to Baseline Visit.

    Participation in clinical trial with biological investigational agents (last study visit occurring) within 90 days prior to Baseline Visit. Participation in any other investigational clinical trial while participating in this clinical trial.
11. Previous participation in any zavegepant study within the last 2 years.
12. ANY of the following findings at the Screening Visit and laboratory tests as assessed by the study-specific laboratory:

    1. Class 2 or Class 3 obesity, defined as body mass index >35 kg/m2.
    2. Estimated Globular Filtration Rate <30 mL/min/1.73 m2.
    3. Total bilirubin ≥1.5 × upper limit of normal.
    4. Liver transaminases ≥2.0 × upper limit of normal .
    5. Neutrophil count ≤1000/μL (or equivalent).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2027-08-02 (Estimated); Study Completion 2027-08-02 (Estimated)

PRIMARY OUTCOMES:
Comparing efficacy of zavegepant with placebo in the acute treatment of migraine as measured by pain freedom at 2-hours post dose during the Double-Blind Treatment (DBT) Phase. | 2 hours post-dose
  Pain levels will be assessed on a 4-point scale (0=none, 1=mild, 2=moderate, 3=severe) using an electronic handheld device. Pain freedom is measured as a pain level of none at 2 hours post-dose.
Consistency of efficacy of zavegepant across multiple attacks in the acute treatment of migraine as measured by pain freedom at 2-hours post dose during the DBT Phase. | 2 hours post-dose
  Freedom from pain response, defined as pain freedom at 2 hours post-dose in ≥2 of 3 qualifying migraine attacks of moderate to severe in intensity.

SECONDARY OUTCOMES:
Percentage of participants with freedom from Most Bothersome Symptoms (MBS) at 2 hours post-dose | 2 hours post-dose
  Freedom from MBS is defined as the absence of the reported MBS.
Percentage of participants with pain relief at 2 hours post-dose | 2 hours post-dose
  Pain relief is defined as intensity of none or mild.
Percentage of participants with pain relief at 15 minutes post-dose | 15 minutes
  Pain relief is defined as intensity of none or mild.
Percentage of participants with consistency of pain relief for at least 2 of 3 qualifying attacks at 2 hours post-dose | 2 hours post-dose
  Pain relief is defined as intensity of none or mild.
Percentage of participants with return to normal function at 2 hours post-dose | 2 hours post-dose
  Return to normal function is defined as have a functional status of normal.
Percentage of participants with return to normal function at 30 minutes post-dose | 30 minutes post-dose
  Return to normal function is defined as have a functional status of normal.
Percentage of participants with sustained pain freedom from 2 to 48 hours post-dose | 2 to 48 hours post-dose
  Pain freedom is measured as a pain level of none. This outcomes measures pain freedom for the duration of 2 to 48 hours post-dose.
Percentage of participants in the triptan resistant/refractory (TRR) group with pain freedom at the 2 hours post-dose | 2 hours post-dose
  TRR participants are those that have had inadequate responses from at least 2 different triptans as determined by the principal investigator. Pain freedom is measured as a pain level of none.
Percentage of participants with adverse events (AEs) of moderate or severe intensity | Duration of study (up to 26 weeks from signing of the inform consent to the safety follow-up period.
Percentage of participants with serious adverse events (SAEs) | Duration of study (up to 26 weeks from signing of the inform consent to the safety follow-up period.
Percentage of participants with local irritation AEs | Duration of study (up to 26 weeks from signing of the inform consent to the safety follow-up period.
Percentage of participants with grade 3 or 4 laboratory test abnormalities | Duration of study (up to 26 weeks from signing of the inform consent to the safety follow-up period.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C5301007